CLINICAL TRIAL: NCT02779062
Title: ALTE Study: Interviews With Parents of Infants Seen in an Emergency Department
Brief Title: Apparent Life Threatening Events in Infants
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14030
Record Dates: First submitted 2016-04-25; First posted 2016-05-20 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: ALTE
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Interview — Interview

SUMMARY:
Infants sometimes experience sudden symptoms such as breathing irregularities or limpness that frighten parents and prompt them to seek emergency medical care. While few of these episodes are truly life-threatening and require hospital admission, some parents may have been so frightened that they will resist returning home from the emergency department with their baby even if the objective risk is extremely small. Study subjects (parents of infants with an apparent life threatening event) will be contacted and interviewed. Investigators want to learn whether or not study subjects would accept returning home after a brief period of observation in the emergency department if the physician determines that it is safe to do so.

DETAILED DESCRIPTION:
An apparent life-threatening event (ALTE) refers to the sudden occurrence in an infant of symptoms such as breathing irregularities, stiffness, or limpness, that appear frightening to caretakers, prompting them to seek medical care. ALTE was first defined in 1986 by an NIH consensus panel. Population-based epidemiologic studies have reported a range of 2.5 to 9.4 ALTE admissions per 1000 live births.

While few ALTEs are truly life-threatening, both clinicians and parents may assume that the infant's life was-and may still be-in danger until proven otherwise. Since the actual risk of an adverse outcome in a well-appearing ALTE patient is unknown, this concern often leads to an extensive diagnostic evaluation and hospitalization to rule out serious occult pathology even when a patient appears well on presentation and has an unremarkable clinical assessment.

Nonspecific inpatient diagnostic evaluations can harm patients by causing complications from invasive testing, false-positive test results, and vulnerable child syndrome. Given these risks and the low probability that such testing will identify a treatable diagnosis in a well-appearing infant, the American Academy of Pediatrics has established a Guideline Committee on ALTEs to develop recommendations for the management of these patients. Specifically, the Committee is formulating criteria to define a low-risk group of infants presenting with ALTE who may be safely discharged after minimal diagnostic testing and a few hours of observation. While an evidence-based clinical guideline has the potential to reduce unnecessary testing and hospital admissions, anecdotal evidence suggests that some parents may have been so frightened by the event that they will resist returning home with their baby even if the objective risk is extremely small. To gather data about parental attitudes, the investigators propose to survey subjects (parents of infants who have experienced an ALTE) to learn whether or not they would accept returning home after a brief period of observation in the emergency department if the physician determines that it is safe to do so. This survey will focus on subject's willingness to forgo admission to the hospital when the risks associated with hospitalization (e.g., hospital-acquired infection, complications of invasive diagnostic procedures) might outweigh the risk of a recurrent ALTE or serious underlying condition. Subject's with an obvious need for admission based on the initial clinical assessment will be excluded, since discharge home would not be an option. Study findings will inform efforts to develop clinical guidelines for the management of an ALTE that take into account both parental attitudes and objective evidence. Without both types of data, implementation of such a guideline will be problematic.

ELIGIBILITY:
Inclusion Criteria:

* Adult parents of an infant with an ALTE event

Exclusion Criteria:

* Unwilling to sign informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult parents of infants with an apparent life threatening event
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Parental comfort level with disposition home from emergency department | Subject will be asked to describe their experiences in the ER when their infant was undergoing an evaluation following an apparent life-threatening event. Subject will be interviewed face-to-face or by telephone within 3 years of the event.
  Subject response (yes or no) to the following question: Would you have felt comfortable returning home from the emergency department with your baby (rather than admitting baby to the hospital overnight) if the medical evaluation in the emergency department had determined that it would be safe to do so? This question will be asked within the context of a series of questions addressing the subject's experience following the apparent life-threatening event of their infant.

CONTACTS AND LOCATIONS:
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States